CLINICAL TRIAL: NCT04582877
Title: Pressure Guidewire System Multi-center, Prospective, Self-Control, Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zurich Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: WXYL-LC-2018001
Record Dates: First submitted 2020-09-17; First posted 2020-10-12 (Actual); Results first posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- FFR Measurement in Intermediate-Grade Coronary Stenosis (Other): Participants with intermediate-grade coronary stenosis undergo measurement of fractional flow reserve using the test article (Zurich Pressure Guidewire System) and predicate article (Abbott PressureWire System).
  Interventions: Device: FFR measurement

INTERVENTIONS:
Device: FFR measurement — FFR is measured sequentially with the test article and the predicate device.

SUMMARY:
Patients with intermediate-grade coronary stenosis undergo measurement of fractional flow reserve using the test article (Zurich Pressure Guidewire System) and predicate article (Abbott PressureWire System). Both articles are used within the same participant and the FFR values are statistically compared with each other.

DETAILED DESCRIPTION:
The objective of the 'Pressure guidewire system multi-center, prospective, single-subject design clinical trial' is to evaluate the effectiveness and safety of Zurich Medical's pressure guidewire system (including guidewire with high-fidelity sensors and a unique paired portable display unit), which is used to measure the coronary artery blood fractional flow reserve (FFR) to diagnose coronary artery disease, and to direct a catheter through a blood vessel. This clinical trial uses a multi-center, prospective, single-subject design trial method, using St. Jude Medical's pressure guidewire and Analyzer Express as a control device. The subjects who met the criteria for this study will be registered with the central registration system after enrollment. Participants with intermediate-grade coronary stenosis undergo measurement of fractional flow reserve using the test article (Zurich Pressure Guidewire System) and predicate article (Abbott PressureWire System). Both articles are used within the same participant and the FFR values are statistically compared with each other. The subject's FFR of coronary artery stenosis will first be measured using investigational device and recorded, and then measured using control device and recorded. The safety follow-up period is 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years old, gender-unrestricted, non-pregnant female;
* Understand and be willing to sign an informed consent form;
* Diagnosed with coronary heart disease;
* Intrusive ICA and FFR measurement are needed;
* Visual coronary angiography showed at least one moderate stenosis lesion (diameter stenosis of 30% - 70%) on the coronary artery with diameter ≥ 2.5mm

Exclusion Criteria:

* Patient who do not understand or are unwilling to sign an informed consent form;
* Has a history of myocardial infarction;
* Patient with other serious diseases are not suitable for clinical trials, such as a complex congenital heart disease history, severe heart failure(NYHA cardiac function level IV), long QT syndrome, severe hypertension, Severe asthma, severe chronic obstructive pulmonary disease, liver and kidney dysfunction and other serious infections and critical illnesses;
* Coronary intervention surgery contraindications;
* Patient with ATP contraindications (ATP contraindications: sinus syndrome, sinus insufficiency and the elderly with cautious use or no use);
* The clinical manifestations of patients show acute instability, including acute chest pain (sudden appearance), cardiogenic shock, unstable blood pressure (systolic pressure less than 90mmHg), severe congestive heart failure or acute pulmonary edema;
* The angiography shown or suspect of thrombosis;
* The angiography shown or suspect of dissection;
* Left main coronary artery disease, target blood vessels with severe curvature or calcification lesions, total occlusion;
* There are any other factors that the investigator considers unsuitable for inclusion or completion of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, MD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FFR Measurement in Intermediate-Grade Coronary Stenosis
Started | 300
Completed | 292
Not Completed | 8
Not completed — Did not use device measurement | 5
Not completed — No fractional flow reserve test results | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: The study started with 300 participants, however, 7 patients never completed the study. Additionally, 1 participant violated protocol, however, their baseline characteristics were still recorded.
Arm/Group | FFR Measurement in Intermediate-Grade Coronary Stenosis
Number analyzed (Participants) | 293
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.47 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 190
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han | 292
  Other | 1
Region of Enrollment [Number; unit: participants]
  China | 293
Weight [Mean (Standard Deviation); unit: kg] | 68.79 (11.09)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: The Body Mass Index of 9 participants could not be measured.
  kg/m^2
    number analyzed (Participants) | 284
    (all) | 25.04 (3.11)
History of Allergies [Count of Participants; unit: Participants]
  No Allergies | 251
  Yes Allergies | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Diagnostic Consistency When Comparing FFR Measurement Between Control Device and Investigational Device
Description: Diagnostic consistency rate: When the measurement of control device is positive (FFRPW ≤ 0.80) or negative (FFRPW > 0.80), investigational device is also positive (FFRWS ≤ 0.80) or negative (FFRWS > 0.80).
  Each subject will be considered a research unit (for patients with multiple lesions, the method of converting the results of multiple lesions into patient level is defined in the statistical analysis plan), and the coronary artery FFRPW measured by control device will be taken as reference.
  Measurements are taken on patients with both the trial device and control device, sequentially during the same visit.
Time Frame: Acute - all measurements are taken and assessed during each procedure. Each participant completes their procedure in one visit, with each procedure taking up to 30 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | FFR Measurement in Intermediate-Grade Coronary Stenosis
Number analyzed (Participants) | 292
Participants | 274

2. Secondary Outcome: The Sensitivity of the Trial Device Compared to the Control Device in Diagnosing Coronary Heart Disease
Description: After all subjects complete their procedures, using the subjects as the research unit, with the control device's determined coronary artery FFRpw as a reference, and with FFRpw ≤ 0.80 as a positive threshold, the sensitivity of diagnosing coronary heart disease using the trial device is calculated. Sensitivity = Number of subjects with FFRws (≤0.80) / Number of subjects with FFRpw (≤0.80).
  Measurements are taken on patients with both the trial device and control device, sequentially during the same visit.
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of sensitivity
Arm/Group | FFR Measurement in Intermediate-Grade Coronary Stenosis
Number analyzed (Participants) | 292
percentage of sensitivity
  asymptotic normal method | 89.2 [80.9 to 97.5]
  exact probability method | 89.2 [79.1 to 95.6]

3. Secondary Outcome: The Specificity of the Trial Device Compared to the Control Device in Diagnosing Coronary Heart Disease
Description: After all subjects complete their procedures, using the subjects as the research unit, with the control device's determined coronary artery FFRpw as a reference, and with FFRpw ≤ 0.80 as a positive threshold, the specificity of diagnosing coronary heart disease using the trial device is calculated. Specificity = Number of subjects with FFRws (>0.80) / Number of subjects with FFRpw (>0.80).
  Measurements are taken on patients with both the trial device and control device, sequentially during the same visit.
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of specificity
Arm/Group | FFR Measurement in Intermediate-Grade Coronary Stenosis
Number analyzed (Participants) | 292
Percentage of specificity
  asymptotic normal method | 95.2 [92.1 to 98.2]
  exact probability method | 95.2 [91.5 to 97.6]

4. Secondary Outcome: Positive Predictive Value (PPV) of the Trial Device for Diagnosing Coronary Heart Disease
Description: using the subjects as the research unit, with the control device's determined coronary artery FFRpw as a reference, and with FFRpw ≤ 0.8 as a positive threshold, the positive predictive value of diagnosing coronary heart disease using the trial device is calculated.
  PPV = true positive / (true positive + false positive)
  Measurements are taken on patients with both the trial device and control device, sequentially during the same visit.
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of PPV
Arm/Group | FFR Measurement in Intermediate-Grade Coronary Stenosis
Number analyzed (Participants) | 292
Percentage of PPV
  asymptotic normal method | 84.1 [74.7 to 93.4]
  exact probability method | 84.1 [73.3 to 91.8]

5. Secondary Outcome: Negative Predictive Value (NPV) of the Trial Device for Diagnosing Coronary Heart Disease
Description: After all subjects complete their procedures, using the subjects as the research unit, with the control device's determined coronary artery FFRpw as a reference, and with FFRpw ≤ 0.8 as a positive threshold, the negative predictive value of diagnosing coronary heart disease using the trial device is calculated.
  NPV = true negative / (true negative + false negative)
  Measurements are taken on patients with both the trial device and control device, sequentially during the same visit.
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of NPV
Arm/Group | FFR Measurement in Intermediate-Grade Coronary Stenosis
Number analyzed (Participants) | 292
Percentage of NPV
  asymptotic normal method | 96.9 [94.3 to 99.4]
  exact probability method | 96.9 [93.6 to 98.7]

6. Secondary Outcome: Receiver Operating Characteristic (ROC) Curve of the Trial Device in Diagnosing Coronary Heart Disease
Description: On a two-dimensional coordinate graph, set the x-axis as the false positive rate (FPR), and the y-axis as the true positive rate (TPR). For the FFRws values measured by the trial device, a point pair of TPR and FPR can be obtained based on its performance on the test sample. Adjust the diagnostic threshold of FFRws to obtain a series of points, connect them in sequence (including the points (0,0) and (1,1)), which forms the ROC curve of FFRws. The value of Area Under Curve (AUC) is the size of the area under the ROC curve. The curve is plotted using MedCalc software.
  Measurements are taken on patients with both the trial device and control device, sequentially during the same visit.
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion Probability
Arm/Group | FFR Measurement in Intermediate-Grade Coronary Stenosis
Number analyzed (Participants) | 292
Proportion Probability | 0.9511 [0.92 to 0.98]

7. Secondary Outcome: Passing-Bablok Regression Analysis Results for the Trial Device in Diagnosing Coronary Heart Disease
Description: Using the vessel as the research unit, with the trial device's measured coronary artery FFRws value as the y-axis, and the control device's measured coronary FFRpw value as the x-axis, perform linear regression analysis on the FFR measurement results, and record the regression analysis equation, slope, and intercept. The analysis will be conducted at the lesion level.
  Regression analysis equation: Y=aX + b
  Measurements are taken on patients with both the trial device and control device, sequentially during the same visit.
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: trial device FFRws/control device FFRpw
Arm/Group | FFR Measurement in Intermediate-Grade Coronary Stenosis
Number analyzed (Participants) | 292
trial device FFRws/control device FFRpw | 1 [0.95 to 1]

8. Secondary Outcome: Bland-Altman Bias Analysis Results for the Trial Device in Diagnosing Coronary Heart Disease
Description: Bland-Altman analysis is a statistical method for evaluating the agreement between two measurement methods and for assessing bias.
  Using the vessel as the research unit, analyze the trial device's measured coronary artery FFRws value and the control device's measured coronary artery FFRpw value using Bland-Altman analysis, and plot the bias graph. Measurements are taken on patients with both the trial device and control device, sequentially during the same visit.
  In the two-dimensional Cartesian coordinate of the bias graph, the x-axis represents the average value of the FFR measured by the two devices for each diseased vessel, and the y-axis represents the difference between the FFR values determined by the two devices for each diseased vessel.
  mean: (x-axis): (FFRws+FFRpw) / 2 absolute error (y-axis): FFRws - FFRpw
  The mean absolute error can then be calculated by taking the average of all absolute errors.
Time Frame: as for outcome 1
Population: Measurements are taken on the same, single Arm/Group with both the trial device as well as the control device. That is, the FFRws and FFRpw are both obtained on the same patient - patients are not separated into groups based on whether the trial device or control device was used. Additionally, the final outcome measure is not intended to report the FFRws and FFRpw values, but to evaluate the agreement between the two measurements using the graph.
Measure: Mean (Standard Deviation); unit: mean absolute error
Arm/Group | FFR Measurement in Intermediate-Grade Coronary Stenosis
Number analyzed (Participants) | 292
mean absolute error | -0.01 (0.03)

9. Secondary Outcome: Pearson Linear Correlation Analysis Results for the Trial Device in Diagnosing Coronary Heart Disease
Description: After all subjects complete their procedures, using the vessel as the research unit, perform Pearson linear correlation analysis on the trial device's measured coronary artery FFRws value and the control device's measured coronary artery FFRpw value, and record the correlation coefficient.
  The correlation coefficient is a statistical measure that determines the strength of a linear relationship between two variables, ranging from -1 to 1. A value close to 1 represents a strong positive correlation between the x and y axis values (trail device FFRws and control device FFRpw). Because of the nature of this value, the measure type is "number".
  The coefficient is determined using the following formula:
  P = Cov(x,y) / OxOy
  where: Cov(x,y) = covariance of variables x and y Ox = standard deviation of x Oy = standard deviation of y
Time Frame: as for outcome 1
Measure: Number; unit: Correlation Coefficient
Arm/Group | FFR Measurement in Intermediate-Grade Coronary Stenosis
Number analyzed (Participants) | 292
Correlation Coefficient | 0.9091

10. Secondary Outcome: Device Success Rate Analysis Results for Subjects
Description: After all subjects complete their procedures, using the vessel as the research unit, with valid FFRws and FFRpw readings as the standard for successful device use, compare the device success rates of the trial device and the control device. Success rate is determined as the number of units that were performed successfully on the patient. The case was deemed successful if the unit was able to read a valid FFRws and FFRpw reading.
  Measurements are taken on patients with both the trial device and control device, sequentially during the same visit.
Time Frame: as for outcome 1
Measure: Number; unit: Number of successful devices
Groups:
- FFR Measurement in Intermediate-Grade Coronary Stenosis - Test Article: Participants with intermediate-grade coronary stenosis undergo measurement of fractional flow reserve using the test article (Zurich Pressure Guidewire System).
  FFR measurement: FFR is measured sequentially with the test article and the predicate device.
- FFR Measurement in Intermediate-Grade Coronary Stenosis - Predicate Article: Participants with intermediate-grade coronary stenosis undergo measurement of fractional flow reserve using the predicate article (Abbott PressureWire System).
  FFR measurement: FFR is measured sequentially with the test article and the predicate device.
Arm/Group | FFR Measurement in Intermediate-Grade Coronary Stenosis - Test Article | FFR Measurement in Intermediate-Grade Coronary Stenosis - Predicate Article
Number analyzed (Participants) | 293 | 293
Number of successful devices | 292 | 293

ADVERSE EVENTS:
Time Frame: Acute - following an initial screening visit, each participant completes their procedure in one visit, with each procedure taking up to 30 minutes. Follow-up time is 48 hours post-operatively. Adverse event data can be collected during the day of the procedure, or up to 48 hours afterwards during the follow up period (Visit 3). During the follow-up period, laboratory tests are performed to check for adverse events, comparing blood and other biochemical changes before and after surgery.
Groups:
- FFR Measurement in Intermediate-Grade Coronary Stenosis - Subject Device: Participants with intermediate-grade coronary stenosis undergo measurement of fractional flow reserve using the test article (Zurich Pressure Guidewire System).
  FFR measurement: FFR is measured sequentially with the test article and the predicate device.
- FFR Measurement in Intermediate-Grade Coronary Stenosis - Control Device: Participants with intermediate-grade coronary stenosis undergo measurement of fractional flow reserve using the predicate article (Abbott PressureWire System).
  FFR measurement: FFR is measured sequentially with the test article and the predicate device.
Arm/Group | FFR Measurement in Intermediate-Grade Coronary Stenosis - Subject Device | FFR Measurement in Intermediate-Grade Coronary Stenosis - Control Device
All-Cause Mortality (participants affected / at risk) | 0/295 | 0/295
Serious Adverse Events (participants affected / at risk) | 0/295 | 0/295
Other Adverse Events (participants affected / at risk) | 1/295 | 0/295
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FFR Measurement in Intermediate-Grade Coronary Stenosis - Subject Device (N=295) | FFR Measurement in Intermediate-Grade Coronary Stenosis - Control Device (N=295)
Myocardial injury (Surgical and medical procedures) | 1 | 0 — perioperative

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT04582877/Prot_SAP_001.pdf